CLINICAL TRIAL: NCT01430936
Title: Remote Monitoring of Heart Failure Patients (REMOTE-HF-1) Study - to Assess Utility of a Mobile Device for Improved Management of At-risk Patients
Brief Title: Evaluate Heart Failure Patients With Specially Designed Patient Adherence and Monitoring Software on Standard Mobile Devices
Acronym: REMOTE-HF-1
Status: Completed | Type: Observational
Sponsor: Aventyn, Inc. (Industry)
Collaborators: AT&T (Unknown); BMS Hospital Trust (Other); University of California (Other); Zephyr Technology (Other)
Responsible Party: Sponsor
Other Study IDs: AVN-111
Record Dates: First submitted 2011-08-12; First posted 2011-09-09 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-07

CONDITIONS: Cardiac Decompensation
Keywords: Vascular Diseases; Hypertension; Chronic Kidney Disease; COPD
MeSH Terms: conditions — Heart Failure; Vascular Diseases; Hypertension; Renal Insufficiency, Chronic; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is planned as a feasibility study. The objective is to evaluate a specially designed patient adherence and monitoring software on standard mobile devices in remote monitoring of heart failure patients.

DETAILED DESCRIPTION:
Heart failure is a common cardiovascular problem which is increasing in both prevalence and incidence and associated with substantial morbidity and mortality. The management of heart failure patients is complex and has become a priority world over. Effective methods to keep heart failure patients out of the hospital are essential, both in the interests of the patient's health, as well as to reduce the burden on the health care system.

Heart failure patients should be in a position to provide readings of their weight, blood pressure, fluid intake, medications and other important parameters and communicate this data to care providers using wireless technology. This data should be made available to medical personnel regularly and on a periodic basis. In this manner the health care providers can detect and respond to warning signs or alerts before the patient's condition worsens to warrant a visit to the doctor or a hospital admission with features of heart failure decompensation.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of either gender above the age of 18 years
* The subject is able and willing to provide written informed consent prior to enrollment in the study
* New York Heart Association (NYHA) classification class of II-IV
* Left ventricular ejection fraction (LVEF) less than 40%
* One or more prior hospitalization within the last six months for symptoms, management of heart failure.

Exclusion Criteria:

* Disability of fingers or upper limbs (unable to use devices)
* Visually impaired
* Those unable to read and write
* Hearing dysfunction
* Significant cognitive disabilities, mental illness
* Those who are unable to handle electronic devices
* Those residing in places outside the local mobile phone coverage
* Chronic renal failure on renal replacement therapy
* Patients who may not come for follow up or likely to drop out of the study
* Those awaiting cardiac transplantation
* Any illness which may preclude regular follow up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Tertiary care population
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2011-01; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Measuring resiliency and reliability of mobile technology for transmitting and retrieval of daily patient vital signs and symptoms as per discharge guideline | 3 months
  Investigators instruct patients to send the clinical data (all measured parameters plus symptoms experienced over the previous 24 hours) via the mobile device every day to the local investigator. The monitoring site maintains a log of all data transmitted and received from the patient and to the patient and, any device malfunction/technical problems, unscheduled SMS/Text messages from patient and to the patient is also to be documented in the case report form for the entire duration of study.

SECONDARY OUTCOMES:
Measuring quality of life score of heart failure patients on a qualitative scale | 3 Months

CONTACTS AND LOCATIONS:
Overall Officials: Satish C Govind, MD, PhD, Principal Investigator — Vivus-BMJ Heart Centre; Marcus Stahlberg, MD, PhD, Principal Investigator — Karolinska University Hospital; Bagirath K, MD, Study Director — Narayana Hruduyalaya Hospital; Justine S Lachmann, MD, Study Director — Winthrop University Hospital; Nicole Orr, MD, Study Director — Saint Francis Hospital
Locations (5):
- United States (2):
  - Winthrop University Hospital, Mineola, New York
  - Saint Francis Hospital, Roslyn, New York
- India (2):
  - Narayana Hrudayalaya Hospital, Bangalore, Karnataka
  - Vivus-BMJ Heart Centre, Bangalore, Karnataka
- Karolinska University Hospital, Stockholm, Stockholm County, Sweden

REFERENCES:
- [Background] Hunt SA, Abraham WT, Chin MH, Feldman AM, Francis GS, Ganiats TG, Jessup M, Konstam MA, Mancini DM, Michl K, Oates JA, Rahko PS, Silver MA, Stevenson LW, Yancy CW, Antman EM, Smith SC Jr, Adams CD, Anderson JL, Faxon DP, Fuster V, Halperin JL, Hiratzka LF, Jacobs AK, Nishimura R, Ornato JP, Page RL, Riegel B; American College of Cardiology; American Heart Association Task Force on Practice Guidelines; American College of Chest Physicians; International Society for Heart and Lung Transplantation; Heart Rhythm Society. ACC/AHA 2005 Guideline Update for the Diagnosis and Management of Chronic Heart Failure in the Adult: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines (Writing Committee to Update the 2001 Guidelines for the Evaluation and Management of Heart Failure): developed in collaboration with the American College of Chest Physicians and the International Society for Heart and Lung Transplantation: endorsed by the Heart Rhythm Society. Circulation. 2005 Sep 20;112(12):e154-235. doi: 10.1161/CIRCULATIONAHA.105.167586. Epub 2005 Sep 13. No abstract available. PMID 16160202